CLINICAL TRIAL: NCT02837055
Title: Prospective, Randomized Study in Critically Ill Patients Receiving Endotracheal Intubation: Comparison Between a Conventional Approach and Video Assisted Intubation by the VivaSight™-SL Tube
Brief Title: Conventional Intubation Versus VivaSight™-SL
Acronym: VivaITN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VivaITN
Record Dates: First submitted 2016-06-13; First posted 2016-07-19 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Insufficiency
Keywords: intubation, intratracheal; critical care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VivaSight intubation (Experimental): Patients are intubated with the VivaSight-SL endotracheal tube
  Interventions: Device: VivaSight intubation
- conventional intubation (Active Comparator): Patients are intubated with a conventional endotracheal tube
  Interventions: Device: conventional intubation

INTERVENTIONS:
Device: VivaSight intubation — patients are intubated with an endotracheal tube with an integrated camera
  Arms: VivaSight intubation
Device: conventional intubation — patients are intubated with a conventional endotracheal tube
  Arms: conventional intubation

SUMMARY:
It has been shown that videolaryngoscopy may be superior to direct laryngoscopy for endotracheal intubation in intensive care. Recently, an endotracheal tube with an integrated camera at its tip has been introduced (VivaSight-SL) allowing for direct visual confirmation of the tube's passage through the vocal cords during intubation.

Patients who are requiring urgent or endotracheal intubation in intensive care are randomized to receive either a conventional intubation with direct laryngoscopy or to receive intubation with the VivaSight-SL-Tube. Primary outcome measures are first attempt success rate and number of attempts to successful intubation.

DETAILED DESCRIPTION:
Background

Airway management in critically ill patients is usually performed by endotracheal intubation with direct laryngoscopy. [1, 2] However, it has been shown that videolaryngoscopy may be superior to the conventional approach in intensive care, i. e. the number of attempts to successful intubation and the rate of accidental esophageal intubation are lower and the visualization of the vocal chords is improved. [3, 4]

Recently, an endotracheal tube with an integrated camera at its tip has been introduced that permits a continuous visualization of the tube's insertion into the trachea on a monitor connected to the camera (VivaSightTM-SL, ETView Ltd., Misgav, Israel) [5]. This tube has been CE and FDA certified (http://www.etview.com/products/vivasight-sl).

It is possible to observe the passage of the tube through the vocal chords during intubation and to verify the correct placement by visualization of the tracheal cartilage. This is an advantage over videolaryngoscopy, in which the camera is mounted on the laryngoscope blade. For the VivaSightTM-SL tube, a decrease for time to intubation and an increase of first attempt success has been shown over conventional intubation in a simulator trial. [6]

In this study, the VivaSightTM-SL tube is tested against the conventional approach during elective and urgent intubations in critically ill patients.

Methods

Study design: randomized, prospective trial

Sample size: n = 54

With a sample size of 54 (randomized 1:1 as 2x 27) a difference of 35% for first attempt success over conventional intubation may be detected with an α-error of 0,05 and a β-error of 1-0,8.

Duration of study: until sample size reached or 18 months after begin of study

Procedures:

* screening of patients for study inclusion according to inclusion and exclusion criteria
* conventional endotracheal intubation by direct laryngoscopy
* endotracheal intubation with the VivaSightTM-SL tube

study inclusion:

All patients being treated in the Dept. of Intensive Care Medicine receiving percutaneous tracheotomy due to long term ventilation are screened according to inclusion and exclusion criteria.

Details of study related procedures:

Intubation:

The Intubation with the VivaSightTM-SL endotracheal tube does not differ from an intubation with a conventional tube that is done with respect to the standard operating procedure (SOP) of the Dept. of Intensive Care Medicine. Additionally, the intubation is guided by the camera mounted on the tip of the tube. During the intubation, vital parameters are monitored with respect to the underlying disease and patients' therapy is continuously adjusted. According to the SOP, two physicians are present of which at least one is a fellow or an attending physician with experience in intensive care medicine. In this trial, intubation is done exclusively by a fellow or attending physician.

Consent: all patients or their legal surrogate give written informed consent.

Data protection: Data are anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving urgent or elective endotracheal intubation in the Dept. of Intensive Care Medicine.
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Age < 18 years
* No consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
first attempt success rate | day 1
  after first attempt of intubation
total number of attempts to successful intubation | day 1
  after successful intubation

SECONDARY OUTCOMES:
average number of attempts for intubation | day 1
  after successful intubation
time to successful intubation | day 1
  after successful intubation
time to successful intubation with one attempt | day 1
  after first attempt successful intubation, if applicable
vomiting or aspiration during intubation | day 1
  after successful intubation
accidental esophageal intubation | day 1
  after successful intubation
decrease of SpO2 < 80% | day 1
  after successful intubation, SpO2: oxygen saturation by pulse oximetry
hypotension | day 1
  after successful intubation, hypotension defined as systolic blood pressure < 70mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kluge, MD, PhD, Principal Investigator — Head of Dept. of Intensive Care Medicine
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Braune S, Kluge S. [Airway management]. Dtsch Med Wochenschr. 2014 Oct;139(40):2003-5. doi: 10.1055/s-0034-1387247. Epub 2014 Sep 25. No abstract available. German. PMID 25254395
- [Background] Pothmann W, Kluge S. [Endotracheal intubation]. Dtsch Med Wochenschr. 2010 May;135(3):94-7. doi: 10.1055/s-0029-1244824. Epub 2010 Jan 14. No abstract available. German. PMID 20077384
- [Background] Mosier JM, Whitmore SP, Bloom JW, Snyder LS, Graham LA, Carr GE, Sakles JC. Video laryngoscopy improves intubation success and reduces esophageal intubations compared to direct laryngoscopy in the medical intensive care unit. Crit Care. 2013 Oct 14;17(5):R237. doi: 10.1186/cc13061. PMID 24125064
- [Background] Silverberg MJ, Li N, Acquah SO, Kory PD. Comparison of video laryngoscopy versus direct laryngoscopy during urgent endotracheal intubation: a randomized controlled trial. Crit Care Med. 2015 Mar;43(3):636-41. doi: 10.1097/CCM.0000000000000751. PMID 25479112
- [Background] Huitink JM, Koopman EM, Bouwman RA, Craenen A, Verwoert M, Krage R, Visser IE, Erwteman M, van Groeningen D, Tijink R, Schauer A. Tracheal intubation with a camera embedded in the tube tip (Vivasight() ). Anaesthesia. 2013 Jan;68(1):74-8. doi: 10.1111/anae.12065. Epub 2012 Nov 5. PMID 23121322
- [Background] Kurowski A, Szarpak L, Truszewski Z, Czyzewski L. Can the ETView VivaSight SL Rival Conventional Intubation Using the Macintosh Laryngoscope During Adult Resuscitation by Novice Physicians?: A Randomized Crossover Manikin Study. Medicine (Baltimore). 2015 May;94(21):e850. doi: 10.1097/MD.0000000000000850. PMID 26020389
- [Derived] Grensemann J, Eichler L, Wang N, Jarczak D, Simon M, Kluge S. Endotracheal tube-mounted camera-assisted intubation versus conventional intubation in intensive care: a prospective, randomised trial (VivaITN). Crit Care. 2018 Sep 22;22(1):235. doi: 10.1186/s13054-018-2152-4. PMID 30241488